CLINICAL TRIAL: NCT07245667
Title: Clinical Study to Assess Tolnaftate 1% With a Novel Vehicle for the Treatment of Tinea Pedis
Brief Title: Topical Tolnaftate Stick for Tinea Pedis: An Open-Label Interventional Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Propedix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO-TP-001
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Tinea Pedis
Keywords: tinea pedis; athletes foot
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tolnaftate Stick Formula A (Experimental): Participants will receive Formula A, a topical 1% tolnaftate formulation delivered through a stick-based applicator. The product is applied twice daily for four weeks.
  Interventions: Drug: 1% Tolnaftate Stick Formula A
- Tolnaftate Stick Formula B (Experimental): Participants will receive Formula B, a topical 1% tolnaftate formulation delivered through a stick-based applicator. The product is applied twice daily for four weeks.
  Interventions: Drug: 1% Tolnaftate Stick Formula B
- Tolnaftate Stick Formula C (Experimental): Topical antifungal stick containing 1% tolnaftate in the Formula C base. Applied twice daily for 4 weeks.
  Interventions: Drug: 1% Tolnaftate Stick Formula C

INTERVENTIONS:
Drug: 1% Tolnaftate Stick Formula A — Topical antifungal stick containing 1% tolnaftate in the Formula A base. Applied twice daily for 4 weeks.
  Arms: Tolnaftate Stick Formula A
Drug: 1% Tolnaftate Stick Formula B — Topical antifungal stick containing 1% tolnaftate in the Formula B base. Applied twice daily for 4 weeks.
  Arms: Tolnaftate Stick Formula B
Drug: 1% Tolnaftate Stick Formula C — Topical antifungal stick containing 1% tolnaftate in the PP2C-2003 base formulation. Applied twice daily for 30 days.
  Arms: Tolnaftate Stick Formula C

SUMMARY:
This study is designed to evaluate the safety and effectiveness of multiple 1% tolnaftate formulations delivered through novel stick-based vehicles in individuals with tinea pedis (athlete's foot).

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of 1% tolnaftate formulations delivered through novel stick-based vehicles in the treatment of subjects with potassium hydroxide (KOH)-positive tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 16 or above
* Clinical diagnosis of tinea pedis (For Cohort 4, positive symptomology is acceptable)
* Confirmation of diagnosis with positive potassium hydroxide (KOH) microscopy (For Cohort 4, a negative KOH test is acceptable)
* Signed and dated informed consent form
* Willingness to comply with study protocol and availability for the duration of the study

Exclusion Criteria:

* Diagnosis of moccasin-type tinea pedis
* Presence of serous exudate or pus
* Treatment with a topical antifungal in the past 2 weeks
* Treatment with a systemic antifungal in the past 4 weeks
* Concurrent immunosuppressive or antimicrobial therapy
* Liver disease
* Pregnancy or breastfeeding
* Use any other antifungal therapy during trial or within three months of starting the trial
* Known hypersensitivity to any ingredients of trial agents
* Patients with a current diagnosis of diabetes or neuropathy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects with a Complete Cure at Week 4 | Week 4
  Primary Efficacy Endpoint: Effective treatment, defined as mycological cure, based on a negative potassium hydroxide (KOH) test at week 4.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kuchnir Dermatology and Dermatological Surgery, Framingham, Massachusetts
  - Kuchnir Dermatology and Dermatological Surgery, Milford, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the study team because this is a small study designed for internal evaluation of formulation performance and tolerability. Data will be presented only in aggregated, de-identified form in any publications or presentations.